CLINICAL TRIAL: NCT02374567
Title: Pharmacovigilance in Gerontopsychiatric Patients
Acronym: GAP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAP-2014
Record Dates: First submitted 2015-01-05; First posted 2015-03-02 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Dementia; Depression; Schizophrenia; Psychosomatic Disorders; Anxiety Disorders
Keywords: geriatric psychiatry; pharmacovigilance
MeSH Terms: conditions — Dementia; Depression; Schizophrenia; Psychophysiologic Disorders; Anxiety Disorders | interventions — Phenobarbital; Phenytoin; Carbamazepine; Oxcarbazepine; Valproic Acid; Lamotrigine; Topiramate; Gabapentin; Levetiracetam; Pregabalin; Lacosamide; Clonazepam; Biperiden; Methotrimeprazine; Fluphenazine; Perphenazine; Perazine; Thioridazine; Haloperidol; metylperon; pipamperone; bromperidol; Benperidol; sertindole; ziprasidone; Flupenthixol; Chlorprothixene; Clopenthixol; Fluspirilene; Pimozide; Clozapine; Olanzapine; Quetiapine Fumarate; Sulpiride; Tiapride Hydrochloride; Amisulpride; prothipendyl; Risperidone; Aripiprazole; Paliperidone Palmitate; Diazepam; Oxazepam; Lorazepam; Bromazepam; Clobazam; Alprazolam; Hydroxyzine; Buspirone; Chloral Hydrate; Flurazepam; Nitrazepam; Triazolam; lormetazepam; Temazepam; Midazolam; brotizolam; zopiclone; Zolpidem; zaleplon; Melatonin; Chlormethiazole; Diphenhydramine; Promethazine; Imipramine; Clomipramine; Opipramol; Trimipramine; Amitriptyline; Nortriptyline; Doxepin; Maprotiline; amitriptyline N-oxide; Fluoxetine; Citalopram; Paroxetine; Sertraline; Fluvoxamine; Escitalopram; Tranylcypromine; Moclobemide; Mianserin; Trazodone; Mirtazapine; Bupropion; Venlafaxine Hydrochloride; Reboxetine; Duloxetine Hydrochloride; agomelatine; Pyrithioxin; Piracetam; Donepezil; Rivastigmine; Galantamine; Memantine; Nicergoline; Acamprosate; Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psychiatric drugs (Experimental)
  Interventions: Drug: Phenobarbital; Drug: Phenytoin; Drug: Carbamazepine; Drug: Oxcarbazepine; Drug: Valproic Acid; Drug: Lamotrigine; Drug: Topiramate; Drug: Gabapentin; Drug: Levetiracetam; Drug: Pregabalin; Drug: Lacosamide; Drug: Clonazepam; Drug: Biperiden; Drug: Levomepromazine; Drug: Fluphenazine; Drug: Perphenazine; Drug: Perazine; Drug: Thioridazine; Drug: Haloperidol; Drug: Melperone; Drug: Pipamperone; Drug: Bromperidol; Drug: Benperidol; Drug: Sertindole; Drug: Ziprasidone; Drug: Flupentixol; Drug: Chlorprothixene; Drug: Zuclopenthixol; Drug: Fluspirilene; Drug: Pimozide; Drug: Clozapine; Drug: Olanzapine; Drug: Quetiapine; Drug: Sulpiride; Drug: Tiapride; Drug: Amisulpride; Drug: Prothipendyl; Drug: Risperidone; Drug: Aripiprazole; Drug: Paliperidone; Drug: Diazepam; Drug: Oxazepam; Drug: Lorazepam; Drug: Bromazepam; Drug: Clobazam; Drug: Alprazolam; Drug: Hydroxyzine; Drug: Buspirone; Drug: Chloral Hydrate; Drug: Flurazepam; Drug: Nitrazepam; Drug: Triazolam; Drug: Lormetazepam; Drug: Temazepam; Drug: Midazolam; Drug: Brotizolam; Drug: Zopiclone; Drug: Zolpidem; Drug: Zaleplon; Drug: Melatonin; Drug: Clomethiazole; Drug: Diphenhydramine; Drug: Promethazine; Drug: Imipramine; Drug: Clomipramine; Drug: Opipramol; Drug: Trimipramine; Drug: Amitriptyline; Drug: Nortriptyline; Drug: Doxepin; Drug: Maprotiline; Drug: Amitriptyline oxide; Drug: Fluoxetine; Drug: Citalopram; Drug: Paroxetine; Drug: Sertraline; Drug: Fluvoxamine; Drug: Escitalopram; Drug: Tranylcypromine; Drug: Moclobemide; Drug: Mianserin; Drug: Trazodone; Drug: Mirtazapine; Drug: Bupropion; Drug: Venlafaxine; Drug: Reboxetine; Drug: Duloxetine; Drug: Agomelatine; Drug: Pyritinol; Drug: Piracetam; Drug: Donepezil; Drug: Rivastigmine; Drug: Galantamine; Drug: Memantine; Drug: Nicergoline; Drug: Acamprosate; Drug: Lithium

INTERVENTIONS:
Drug: Phenobarbital
Drug: Phenytoin
Drug: Carbamazepine
Drug: Oxcarbazepine
Drug: Valproic Acid
Drug: Lamotrigine
Drug: Topiramate
Drug: Gabapentin
Drug: Levetiracetam
Drug: Pregabalin
Drug: Lacosamide
Drug: Clonazepam
Drug: Biperiden
Drug: Levomepromazine
Drug: Fluphenazine
Drug: Perphenazine
Drug: Perazine
Drug: Thioridazine
Drug: Haloperidol
Drug: Melperone
Drug: Pipamperone
Drug: Bromperidol
Drug: Benperidol
Drug: Sertindole
Drug: Ziprasidone
Drug: Flupentixol
Drug: Chlorprothixene
Drug: Zuclopenthixol
Drug: Fluspirilene
Drug: Pimozide
Drug: Clozapine
Drug: Olanzapine
Drug: Quetiapine
Drug: Sulpiride
Drug: Tiapride
Drug: Amisulpride
Drug: Prothipendyl
Drug: Risperidone
Drug: Aripiprazole
Drug: Paliperidone
Drug: Diazepam
Drug: Oxazepam
Drug: Lorazepam
Drug: Bromazepam
Drug: Clobazam
Drug: Alprazolam
Drug: Hydroxyzine
Drug: Buspirone
Drug: Chloral Hydrate
Drug: Flurazepam
Drug: Nitrazepam
Drug: Triazolam
Drug: Lormetazepam
Drug: Temazepam
Drug: Midazolam
Drug: Brotizolam
Drug: Zopiclone
Drug: Zolpidem
Drug: Zaleplon
Drug: Melatonin
Drug: Clomethiazole
Drug: Diphenhydramine
Drug: Promethazine
Drug: Imipramine
Drug: Clomipramine
Drug: Opipramol
Drug: Trimipramine
Drug: Amitriptyline
Drug: Nortriptyline
Drug: Doxepin
Drug: Maprotiline
Drug: Amitriptyline oxide
Drug: Fluoxetine
Drug: Citalopram
Drug: Paroxetine
Drug: Sertraline
Drug: Fluvoxamine
Drug: Escitalopram
Drug: Tranylcypromine
Drug: Moclobemide
Drug: Mianserin
Drug: Trazodone
Drug: Mirtazapine
Drug: Bupropion
Drug: Venlafaxine
Drug: Reboxetine
Drug: Duloxetine
Drug: Agomelatine
Drug: Pyritinol
Drug: Piracetam
Drug: Donepezil
Drug: Rivastigmine
Drug: Galantamine
Drug: Memantine
Drug: Nicergoline
Drug: Acamprosate
Drug: Lithium

SUMMARY:
The purpose of this multicenter-study is to investigate safety of psychopharmacological treatment and rates of adverse drug reactions in gerontopsychiatric inpatients. Elderly people are at higher risk for developing side effects under pharmacological treatment due to an altered metabolic situation, higher comorbidity rates and often polypharmacy. Furthermore gerontopsychiatric patients can often not articulate their symptoms clearly, for example due to pronounced cognitive impairment.

The aim of the study is to gain valid data of possible adverse drug reaction rates, their potential risk factors and outcome, as well as medical prescription practises.

To assess these outcomes an intensive pharmacovigilance-monitoring will be conducted at the five participating study sites.

At Baseline demographic data, previous and present disorders, use of drugs, previous and present medication, quality of life, cognitive function, physical examination results, laboratory results and ECG will be assessed.

Afterwards patients are visited weekly and screened for possible adverse drug reactions. All adverse drug reactions will be coded in the MedDRA-system.

In case of a possible serious adverse drug reaction serum levels of all psychotropic substances applicated will be assessed. Drug combinations will be analysed using an established advanced bioinformatic tool (mediQ). Diagnosis, medication intake and possible adverse drug reactions are documented continually.

2 weeks after discharge from the ward, patients will be contacted by phone to assess catamnestic data.

ELIGIBILITY:
Inclusion Criteria:

* Age 65+ years old
* Inpatients treated at one of the geriatric psychiatry study sites.
* Signed consent form ( Patient and/or legally authorized custodian)

Exclusion Criteria:

* Patients that are incapable to give their informed consent and are not under legally authorized custodianship.
* Parallel participation in another clinical trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 407 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Assessment of frequency and severity of adverse events | Participants will be followed for the duration of hospital stay and the follow-up-visit, an expected average of 6 weeks

SECONDARY OUTCOMES:
Assessment of cognitive functioning | At baseline visit and at the final visit (expected average of hospital stay: 4 weeks)
  Mini mental state examination, intensive care delirium checklist
Quality of life | At baseline visit and at the final visit (expected average of hospital stay: 4 weeks)
  SF-8
Adverse drug reactions | Continuously during hospital stay (expected average of hospital stay: 4 weeks) and at follow-up two weeks after discharge
  Dosage record and treatment emergent symptoms scale (DOTES), geriatric adverse event rating scale (GEARS)
Serum level of substances | 1 day at occurrence of SAR
Electrocardiogram | At baseline visit, at occurrence of SAR and at the final visit (expected average of hospital stay: 4 weeks)
Medication intake | Patients medication intake 2 weeks before hospitalization, continuously during hospital stay (expected average of hospital stay: 4 weeks) and at follow-up two weeks after discharge
  Morisky medication adherence scale (MMAS) and chart review

CONTACTS AND LOCATIONS:
Overall Officials: Helge Frieling, Prof., MD, Principal Investigator — Hannover Medical School
Locations (5):
- Germany (5):
  - Bezirkskrankenhaus Augsburg, Augsburg
  - Krankenhaus Hedwigshöhe, Berlin
  - Hannover Medical School, Hanover
  - Asklepios Fachklinikum Lübben, Lubin
  - Asklepios Fachklinikum Teupitz, Teupitz

IPD SHARING:
Plan to Share IPD: No